CLINICAL TRIAL: NCT02985580
Title: Effects of Blueberry Juice Consumption on Brain Activation and Perfusion in Healthy Older People
Brief Title: Effects of Blueberry Juice Consumption on Cognitive Function in Healthy Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1314/134617
Record Dates: First submitted 2016-09-13; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-09

CONDITIONS: Cognitive Aging
MeSH Terms: interventions — blueberry extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blueberry (Active Comparator): Blueberry concentrate consumed daily for 12 weeks.
  Interventions: Dietary Supplement: Blueberry
- Placebo (Placebo Comparator): Placebo concentrate consumed daily for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blueberry
  Arms: Blueberry
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Blueberries are rich in flavonoids that possess antioxidant and anti-inflammatory properties, which in rodent models are neuro-protective. The risk of developing dementia is reduced in people habitually consuming high flavonoid intakes, but data from human intervention studies is sparse. We therefore investigated whether 12 weeks of blueberry concentrate supplementation improved cognitive function in healthy elderly via increased brain activation and perfusion.

ELIGIBILITY:
Inclusion Criteria:

* aged 60-80y
* Addenbrooke's Cognitive Examination III questionnaire > 88
* Consuming 5 or less portions of fruit per day

Exclusion Criteria:

Addenbrooke's Cognitive Examination III questionnaire < 88 Contraindications for MRI Consuming more than 5 portions of fruit per day

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Brain perfusion | Change from baseline to 12 weeks dietary supplementation
  MRI - arterial spin labelling

SECONDARY OUTCOMES:
Brain activation | Change from baseline to 12 weeks dietary supplementation
  fMRI whilst performing modified Stroop task
Cognitive function tests | Change from baseline to 12 weeks dietary supplementation
  Cogstate battery of tests
Blood biomarkers of inflammation | Change from baseline to 12 weeks dietary supplementation
  CRP, IL6,
Blood biomarkers of oxidative stress | Change from baseline to 12 weeks dietary supplementation
  protein carbonyls, glutathione
Blood biomarkers of neurogenesis | Change from baseline to 12 weeks dietary supplementation
  BDNF

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Bowtell, PhD, Principal Investigator — University of Exeter

IPD SHARING:
Plan to Share IPD: No